CLINICAL TRIAL: NCT06846749
Title: Reduced Calorie Feeds in the Early Management of Ill Severely Malnourished Children: a Phase I Clinical Trial
Brief Title: Slow Introduction of Nutrition for Ill Malnourished Children
Acronym: F50
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Kamuzu University of Health Sciences (Other); The Eleanor Crook Foundation (Unknown); Children's Investment Fund Foundation (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Robert Bandsma, Staff Physician, Division of Gastroenterology, Hepatology and Nutrition, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000081371
Record Dates: First submitted 2025-02-11; First posted 2025-02-26 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Malnutrition, Severe Acute; Malnutrition, Child; Malnutrition, Infant
Keywords: Overfeeding, Refeeding syndrome, Glucose Dysregulation
MeSH Terms: conditions — Severe Acute Malnutrition; Child Nutrition Disorders; Infant Nutrition Disorders; Refeeding Syndrome

STUDY DESIGN:
Intervention Model Description: This is a parallel interventional study model, making use of the Bayesian Continual Reassessment Method to help allocate patients to the different interventional products related to the risk of hypoglycemia compared to F75. The DSMB will be involved in decisions around continuing with a specific interventional product incorporating SAE data.
Masking Description: This is an open label trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- F75 milk feeds (Active Comparator): F-75 nutritional stabilization feed was designed in the 1990s assuming that severely malnourished children with infections are metabolically vulnerable and have a range of micronutrient disturbances. F75 aims to provide 95 kcal/kg/day and was intended to support children through early stabilization when fighting infections and not aimed at weight gain. Once clinically stabilized, on average after 3-5 days, children are transitioned from F75 to ready-to-use therapeutic foods (RUTF) that provide substantially higher amount of protein and calories to promote rapid weight gain.
  Interventions: Dietary Supplement: F75 milk feeds
- F50 milk feeds (Experimental): The F50 feed has been meticulously formulated by Nutriset. The composition is identical to that of F75, with the only distinction being the reduction in calorie content with F50 aiming to provide 63kcal/kg/day. This ensures that the nutritional parameters and essential components remain consistent, while the lower calorie count aligns with the specific requirements of this trial. Once clinically stabilized, on average after 3-5 days, children are transitioned from F50 to RUTF that provide substantially higher amounts of protein and calories to promote rapid weight gain.
  Interventions: Dietary Supplement: F50 milk feeds
- F35 milk feeds (Experimental): The F35 feed has been meticulously formulated by Nutriset. Their composition is identical to that of F75, with the only distinction being the reduction in calorie content with F35 aiming to provide 47kcal/kg/day. This ensures that the nutritional parameters and essential components remain consistent, while the lower calorie count aligns with the specific requirements of this trial. Once clinically stabilized, on average after 3-5 days, children are transitioned from F35 to RUTF that provide substantially higher amounts of protein and calories to promote rapid weight gain.
  Interventions: Dietary Supplement: F35 milk feeds

INTERVENTIONS:
Dietary Supplement: F75 milk feeds — Standard 'F75' (75 kcal/100 ml) 95 kcal/kg/day 12.05 mg/kg/min glucose
  Other Names: Therapeutic Milk
  Arms: F75 milk feeds
Dietary Supplement: F50 milk feeds — Reduced caloric 'F50' (50kcal/100ml) 63 kcal/kg/day 8.03mg/kg/min glucose
  Other Names: Therapeutic Milk
  Arms: F50 milk feeds
Dietary Supplement: F35 milk feeds — Reduced caloric 'F35' (35 kcal/100ml)
  * 47 kcal/kg/day
  * 5.62 mg/kg/min glucose
  Other Names: Therapeutic Milk
  Arms: F35 milk feeds

SUMMARY:
The goal of this clinical trial is to learn if giving lower calorie feeds during the first stage of treatment helps improve survival in severely malnourished children who are ill. The main question it aims to answer is:

Is it safe to feed ill severely malnourished children lower calorie feeds during the early treatment phase?

Researchers will compare two lower calorie feeds (F50 and F35) to the standard feed (F75) to see if they help children recover safely without increasing their risk of low blood sugar (hypoglycemia).

Participants will:

* Receive one of the lower calorie feeds (F50 or F35) or the standard feed (F75) during their hospital stay.
* Be closely monitored for low blood sugar and signs for worsening of clinical symptoms.
* Be treated until they are stable and ready to be fed more calories to help them gain weight.

DETAILED DESCRIPTION:
Malnutrition is a leading cause of death, contributing to nearly 45% of all deaths in children under the age of 5 years worldwide. In its most severe form, severe malnutrition remains prevalent globally affecting more than 45 million children. Severely malnourished children have a strongly increased risk of death from common infectious diseases. Updates in treatment protocols for severe malnutrition have been the most impactful intervention against childhood mortality.

Management of severely malnourished children hospitalized with critical illness is based on guidelines developed by the World Health Organization and consists of three main components: 1. Clinical stabilization 2. Treatment of underlying infections 3. Nutritional rehabilitation. Clinical stabilization includes administration of broad-spectrum antibiotics, fluid resuscitation (if needed) and providing a nutritional stabilization feed that is called 'F75'. F75 was designed in the 1990's assuming that severely malnourished children with infections are metabolically vulnerable and have a range of micronutrient disturbances. F75 aims to provide 95 kcal/kg/day and was not intended for weight gain since, during this initial period, children are actively fighting infections. Once clinically stabilized, on average after 3-5 days, children are transitioned from F75 to ready-to-use therapeutic foods (RUTF) that provide a substantially higher amount of protein and calories to promote rapid weight gain. Some children fail this transition and have to revert back to F75 for a period of time due to clinical deterioration or not tolerating the RUTF. Despite protocolized management of these highly vulnerable patients, mortality rates have remained high over the past decades and reported to range between 10-30%, depending on population, setting and duration of follow up.

Scientific evidence from the last decade has started to reform the approach to care for critically ill children in relation to feeding. Evidence shows that, during severe infection, the body enters a catabolic state, which is critical for immune function and pathogen clearance. Overfeeding during this phase may disrupt essential metabolic processes, including a process of cellular recycling called autophagy, which play a key role in fighting infections. Studies in both high- and low-resource settings have shown that limiting caloric intake in the early days of critical illness may improve clinical outcomes, including reducing the risk of infections and decreasing ICU stay durations.

No clinical trial has examined the optimal caloric intake for ill severely malnourished children in LMIC and the current F75 composition was only based on expert opinion. Our population and treatment settings are substantially different compared to high income settings. Children in LMIC are often wasted to a degree of severity not frequently observed in high resource settings. Severely malnourished children are thought to be at risk of refeeding syndrome, defined as an acute insulin response to rapid refeeding leading to electrolyte imbalances and hypoglycemia. In many LMIC, health resources are scarce and physician and nurse to patient ratios are low. Malnourished children are therefore managed using relatively protocolized but largely non-evidence-based approaches. This has led the World Health Organization (WHO) to press the scientific community to review of current practices. Intravenous fluid administration is often avoided due to the absence of fluid solutions, infusion pumps and lack of resources to monitor fluid intake. Parenteral nutrition is generally not available. Therefore, fluid and nutrition are mainly provided orally or through a nasogastric tube.

We aim to test the safety and tolerability of using lower caloric feeds during the initial clinical stabilization phase of acutely ill severely malnourished children. Reducing caloric intake has been shown to improve clinical outcomes of critically ill children with malnutrition in high resource setting. We propose that applying a similar strategy during the initial stabilization phase will improve survival of critically ill children with malnutrition in low resource settings. However, reducing caloric intake in these children may increase the risk of hypoglycemia. Therefore, we will conduct a randomized phase I clinical trial specifically designed to assess and minimize this risk. The potential benefits on childhood survival renders this trial ethically and clinically justified. Given current data, the use of lower caloric feeds should be evaluated in this vulnerable population. Conducting this safety phase-I trial will be a critical step before proceeding with an efficacy-focused trial powered for mortality.

The F50 and F35 feeds have been meticulously formulated for this trial. Their composition is identical to that of F75, with the only distinction being the reduction in calorie content with F50 aiming to provide 63kcal/kg/day and F35 aiming to provide 47kcal/kg/day. This ensures that the nutritional parameters and essential components remain consistent, while the lower calorie count aligns with the specific requirements of this trial. Once clinically stabilized, on average after 3-5 days, children are transitioned from F50 or F35 to RUTF that provide substantially higher amounts of protein and calories to promote rapid weight gain. This novel trial design will be used to ensure the highest level of safety. Once the optimal and safe reduction in calories is determined, we would be able to perform a large intervention trial whereby the provided feeds (i.e., standard F75 or a reduced calorie feed) can be randomized and tested for efficacy in reducing mortality. This work has the potential to radically change how we manage seriously ill severely malnourished children and reduce the mortality in the most vulnerable children globally.

ELIGIBILITY:
Inclusion Criteria:

* Age - greater than or equal to 6 months to less than 59 months (age range for which WHO guidelines were developed and where children are not expected to be exclusively breastfeeding
* Admitted to hospital with acute, non-traumatic illness and having received a maximum of 2 feeds of F75 at time of enrolment
* Severe malnutrition (WHZ <-3 z-scores of the median WHO growth standards and/or MUAC <115mm)
* Accompanied by care provider able to provide written or witnessed informed consent
* Primary caregiver plans to stay in the study area for the duration of the study
* Having no more than one clinical sign displayed below "Clinical/Lab Feature & Criteria"

Exclusion Criteria:

* Has oedematous malnutrition (excluded for this safety focused trial as fluid accumulation influences weight which is used to calculate required caloric intake)
* Requires immediate cardiac/respiratory resuscitation (chest compressions/ventilation)
* Clinical contraindications for enteral nutrition
* Admission for traumatic or surgical indication
* Weighs <3.5kg
* Presence of terminal illness likely to result in death within 6 months
* Known congenital heart disease
* Have had 2 documented hypoglycaemic events in hospital
* More than one clinical sign displayed below "Clinical/Lab Feature & Criteria"
* Primary caregiver declines to provide informed consent

Clinical/Lab Feature & Criteria Guidelines

Clinical/Lab Feature: Respiratory distress Oxygenation Criteria: "Subcostal in-drawing" or "nasal flaring" or "head-nodding"

Clinical/Lab Feature: Oxygenation Criteria: "Central cyanosis" or SaO2 <90%

Clinical/Lab Feature: Circulation Criteria: Limb temperature gradient or capillary refill >3 seconds

Clinical/Lab Feature: Reduced conscious level Criteria: AVPU < "A"

Clinical/Lab Feature: Rapid pulse Criteria: Heartbeat per min > 180

Clinical/Lab Feature: Severe anemia Criteria: Haemoglobin < 7g/dl

Clinical/Lab Feature: Hypoglycemia Criteria: Blood glucose < 3mmol/L

Clinical/Lab Feature: Abnormal temperature Criteria: Axial temperature <36 or >38oC

Clinical/Lab Feature: Very low MUAC Criteria: MUAC <11cm

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Episodes of moderate hypoglycemia | During the period of F75/F50/F35 provision meaning the stabilization phase which is on average 3 days
  The occurrence of at least one episode of moderate hypoglycemia (less than or equal to 3.0 mmol/l) during the stabilization phase as measured utilizing the Dexcom Continous Glucose Monitoring Device and/or bed-side glucometer (OneTouch).

SECONDARY OUTCOMES:
Serious Adverse Events | During the period of F75/F50/F35 provision meaning the stabilization phase, which is on average 3 days
  The number of severe adverse events between the intervention (F50 and F35) and control (F75) arms. Diagnosis, date and time of onset, outcome severity and relation to the type of feed administration will be established within 24 hours and reported.
Episodes of hypoglycemia or hyperglycemia | During the period of F75/F50/F35 provision meaning the stabilization phase, which is on average 3 days
  The number of episodes of hypoglycemia (less than or equal to 3.0mmol/l) or hyperglycemia (greater than or equal to 10 mmol/l) and glycemic variability between the intervention (F50 and F35) and control (F75) arms. Measurements will be done utilizing the Dexcom Continuous Glucose Monitoring Device and/or bed-side glucometer (OneTouch).
Duration of the stabilization phase | The duration of the stabilization phase which is expected to be on average 3 days following enrolment.
  The duration of the stabilization phase in days - including when the child "failed to transition" between the intervention (F50 and F35) and control (F75) arms.
Failed transition to ready-to-use-therapeutic foods (RUTF). | Transition phase expected to be on average 3 days following start of RUTF
  Return to stabilization feed after attempting to introduce RUTF.
Duration of hospital stay | Study enrolment to discharge, which is on average 7 days
  Length of time spent in hospital for the duration of the study
Volume of feed consumed per day | During the period of the stabilization phase, which is on average 3 days
  Compare the volume of feeds consumed per day in ml/kg body weight for the interventions (F50 and F35) and control (F75) arms.
Change in weight | Admission to clinical stabilization, which is on average 3 days
  Change in weight from admission to clinical stabilization as determined by anthropometric measurements
Loose or watery stools | Study enrolment to discharge, which is on average 7 days
  The number of loose or watery stools per day, using the Bristol Stool Scale.
Vomiting episodes | Study enrolment to discharge, which is on average 7 days
  Number of vomiting episodes per day
Feeds withheld | During the period of the stabilization phase, which is on average 3 days
  Number of feeds withheld from participant
New Infection | Study enrolment to discharge, which is on average 7 days
  New infection onset as defined by positive bacterial cultures
Mortality | Study enrolment to discharge, which is on average 7 days
  Mortality as a number and percentage during hospitalization.

OTHER OUTCOMES:
Glucose response | The duration of the stabilization phase, which is on average 3 days
  Pre and post prandial glucose response
C-reactive protein and white blood cell count and differential | Enrolment
  C-reactive protein and white blood cell count and differential at enrolment as a biochemical marker of infection severity
Venous blood gas, lactate, electrolytes | Day 3 of admission
  Venous blood gas, lactate, electrolytes at day 3 after hospital admission as a biochemical marker of illness severity and refeeding syndrome
Energy expenditure | Day 1 of admission and discharge, which is expected to be on average after 7 days
  Energy expenditure using Indirect Calorimetry at enrolment and day 1 after discharge

CONTACTS AND LOCATIONS:
Locations (2):
- International Centre for Diarrheal Disease Research, Dhaka, Bangladesh
- Queen Elizabeth Central Hospital, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: No
Only SAE's will be shared as individual participant data to the SAE review committee.

REFERENCES:
- [Background] Fivez T, Kerklaan D, Mesotten D, Verbruggen S, Wouters PJ, Vanhorebeek I, Debaveye Y, Vlasselaers D, Desmet L, Casaer MP, Garcia Guerra G, Hanot J, Joffe A, Tibboel D, Joosten K, Van den Berghe G. Early versus Late Parenteral Nutrition in Critically Ill Children. N Engl J Med. 2016 Mar 24;374(12):1111-22. doi: 10.1056/NEJMoa1514762. Epub 2016 Mar 15. PMID 26975590
- [Background] Maitland K, Berkley JA, Shebbe M, Peshu N, English M, Newton CR. Children with severe malnutrition: can those at highest risk of death be identified with the WHO protocol? PLoS Med. 2006 Dec;3(12):e500. doi: 10.1371/journal.pmed.0030500. PMID 17194194
- [Background] Kerac M, Bunn J, Seal A, Thindwa M, Tomkins A, Sadler K, Bahwere P, Collins S. Probiotics and prebiotics for severe acute malnutrition (PRONUT study): a double-blind efficacy randomised controlled trial in Malawi. Lancet. 2009 Jul 11;374(9684):136-44. doi: 10.1016/S0140-6736(09)60884-9. PMID 19595348
- [Background] Hossain M, Chisti MJ, Hossain MI, Mahfuz M, Islam MM, Ahmed T. Efficacy of World Health Organization guideline in facility-based reduction of mortality in severely malnourished children from low and middle income countries: A systematic review and meta-analysis. J Paediatr Child Health. 2017 May;53(5):474-479. doi: 10.1111/jpc.13443. Epub 2017 Jan 4. PMID 28052519
- [Background] Bhutta ZA, Das JK, Rizvi A, Gaffey MF, Walker N, Horton S, Webb P, Lartey A, Black RE; Lancet Nutrition Interventions Review Group, the Maternal and Child Nutrition Study Group. Evidence-based interventions for improvement of maternal and child nutrition: what can be done and at what cost? Lancet. 2013 Aug 3;382(9890):452-477. doi: 10.1016/S0140-6736(13)60996-4. Epub 2013 Jun 6. PMID 23746776
- [Background] Bhutta ZA, Berkley JA, Bandsma RHJ, Kerac M, Trehan I, Briend A. Severe childhood malnutrition. Nat Rev Dis Primers. 2017 Sep 21;3:17067. doi: 10.1038/nrdp.2017.67. PMID 28933421
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- See also: WHO "Levels and trends in child malnutrition" — https://www.who.int/publications/i/item/9789240025257
- See also: WHO "Updates on the management of severe acute malnutrition in infants and children" — http://apps.who.int/iris/bitstream/10665/95584/1/9789241506328_eng.pdf
- See also: Management of severe malnutrition: a manual for physicians and other senior health workers — http://apps.who.int/iris/bitstream/10665/41999/1/a57361.pdf